### **Principal Investigator:**

Timothy S Pardee, M.D., Ph.D.
Section on Hematology and Oncology
Wake Forest University School of Medicine
Medical Center Blvd.
Winston-Salem, NC 27157

### **Co-Investigators:**

Heidi D. Klepin, M.D., M.S.
Section on Hematology and Oncology
Wake Forest University School of Medicine
Medical Center Blvd.
Winston-Salem, NC 27157

Susan Lyerly, P.A.-C.
Section on Hematology and Oncology
Wake Forest University School of Medicine
Medical Center Blvd.
Winston-Salem, NC 27157

Bayard Powell, M.D.
Section Head, Hematology and Oncology
Wake Forest University School of Medicine
Medical Center Blvd.
Winston-Salem, NC 27157

Megan Manuel, N.P.
Section on Hematology and Oncology
Wake Forest University School of Medicine
Medical Center Blvd.
Winston-Salem, NC 27157

Sarah Dralle, N.P.
Section on Hematology and Oncology
Wake Forest University School of Medicine
Medical Center Blvd.
Winston-Salem, NC 27157

### Biostatistician:

Scott Isom, M.S.
Comprehensive Cancer Center
Wake Forest University School of Medicine
Medical Center Blvd.
Winston-Salem, NC 27157

### NCT01869777

Protocol Version Date 07.25.14

### 1.0 Background and Rationale

The acute leukemias in adults are characterized by resistance and poor outcomes. Acute myeloid leukemia (AML) and acute lymphoid leukemia (ALL) are aggressive malignancies that lead to the accumulation of immature myeloid or lymphoid precursors, resulting in progressive marrow failure and death <sup>1</sup>. They affect approximately 19,000 people per year in the United States; despite decades of research, the overall 5-year survival remains a disappointing 30-40% <sup>2-4</sup>. The current treatment is intensive induction chemotherapy followed by consolidation using chemotherapy or a stem cell transplant <sup>2,5</sup>.

Selecting patients for intensive therapy is a major challenge in the acute leukemias.

There are multiple prognostic factors in the acute leukemias that are used to try and select the best candidates for intensive induction therapy. The most powerful single prognostic factor in the acute leukemias is cytogenetics. Using standard karyotyping techniques patients can be divided into 3 prognostic categories; good, intermediate and poor. They are characterized by 5 year overall survival rates of 55%, 24% and 5% respectively 6. Age is also a powerful prognostic factor in the acute leukemias. For patients over 60 with acute leukemia, the prognosis is grave (five-year survival of less than 10%) 7-9. These patients have many co-morbidities and increased resistant disease <sup>2,5</sup>. Both acute leukemias in adulthood disproportionately affect the elderly (median age of onset of 72 and >60 for AML and ALL, respectively) 4,10. The presence of poorrisk cytogenetic factors is increased in elderly patients as well as expression of multi-drug efflux pumps <sup>11-12</sup>. Performance status is another important prognostic factor and the ability to tolerate induction therapy decreases as performance status worsens regardless of age 8. For older patients with poor performance status it is currently acceptable clinical practice to offer only supportive care. In AML this has led some authors to conclude that standard induction chemotherapy should not be offered to elderly patients<sup>13</sup>. In contrast other groups have found a positive clinical impact of standard therapy in older AML patients with increased survival and less time in hospital than those offered only supportive care 14. In order to better help clinicians decide what patients should be offered intensive therapy a number of prognostic scoring systems have been developed<sup>15</sup>. The majority of these systems rely heavily on the cytogenetics of the leukemia and this information is generally not available at the time of diagnosis. An additional prognostic factor that could be easily obtained at the time of diagnosis would a major step forward. In addition to deciding on what initial therapy to give an AML patient there is another major clinical decision point. A nadir marrow is obtained on day 14 following standard induction therapy and if there is significant residual disease a second course of induction is usually attempted. In many cases patients have experienced significant complications by day 14 making additional chemotherapy difficult to safely administer. There are very few studies on what prognostic factors are important when considering a second course of induction therapy. This is further complicated by the lack of rigorously performed studies to establish the predictive power of a positive nadir marrow. An additional prognostic factor that could be easily obtained on day 14 would be of significant help to clinicians.

**Bioimpedance phase angle is prognostic in multiple disease states.** Phase angle is measured by bioimpedance and reflects cell membrane integrity, nutritional status and muscle mass<sup>16</sup>. It has been found to be prognostic in a number of conditions such as end stage renal disease, HIV and COPD<sup>17-19</sup>. Additionally, it is prognostic in multiple tumor types including pancreatic, colorectal, breast and head and neck. In a recent report it was found to be strongly prognostic for patients with hematologic malignancies undergoing allogeneic stem cell transplants<sup>20</sup>. Standardized phase angle measurements are made non-invasively, can be done quickly and reproducibly and with no patient discomfort. Measurements are taken by placing 2

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

electrodes on the hand and 2 on the foot from the same side of the patient. A small voltage is applied between the electrodes and the timing of induced the current is measured. The current is approximately 1000 times lower than the sensitivity of sensory neurons and thus cannot be felt by the patient and has no known biological effect. This study seeks to establish the feasibility and prognostic power of standardized phase angle in acute leukemia patients undergoing intensive induction chemotherapy.

### 2.0 Objectives

- 2.1 To determine the feasibility of obtaining standardized phase angle measurements on patients hospitalized for treatment of newly diagnosed acute leukemia.
- 2.2 To evaluate the association between standardized phase angle measured at the start of therapy and treatment-related outcomes including:

  Primary outcome: Treatment related mortality (defined as 60-day mortality)

  Secondary outcomes: Evaluate the association of the day 14 standardized phase angle and treatment related outcomes, 30-day mortality, length of hospitalization, transfer to intensive care unit during induction, treatment response (14 day bone marrow response, complete remission), receipt of post-remission therapy, overall survival.
- 2.3 An exploratory analysis investigating associations with the primary and secondary outcomes using different ways to categorize the baseline standardized phase angle measurement (obtained on the first day of treatment) and, for AML patients, the standardized phase angle measure obtained just prior to the nadir marrow.

### 3.0 Patient Selection Criteria

### 3.1 Eligible

- 3.11 Hospitalized for newly diagnosed acute leukemia
- 3.12 Receiving induction treatment while hospitalized
- 3.13 Willing and able to provide written informed consent

### 3.2 Ineligible

- 3.21 Presence of a pacemaker or defibrillator.
- 3.22 Patients pregnant at the time of enrollment.
- 3.23 Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients.
- 3.24 Unable/unwilling to follow protocol requirements

### 4.0 Study Design

Eligible patients with newly diagnosed acute leukemia will have phase angle measurements recorded within the first 3 days of treatment. AML patients will have a second phase angle measurement taken within 2 days of the nadir marrow. Whenever possible, measurements will be taken prior to any invasive procedures (bone marrow biopsy, leukophoresis, PICC line placement, etc.). In addition data on pertinent covariates including age, demographic data, tumor biology, white blood cell count, LDH, need of total parental nutrition or placement of a feeding tube and comorbid conditions

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

will be collected. There will be no intervention done as a result of the phase angle measurement. Patients will be followed at routine visits per standard of care for two years or until death.

### 5.0 <u>Data Management</u>

All data will be de-identified and stored in a password protected REDCap database in accordance with HIPAA. Research Electronic Data Capture (REDCap) software is a secure, web-based application designed to support survey creation, survey administration and data capture for research studies. Records to be kept on each subject will include only the data specified in Appendices B, C, D, E and F. Only study personnel will have access to the data.

### 6.0 Registration

Eligible patients must be registered with the CCCWFU Registrar. Following registration, patients should have a baseline phase angle measurement taken. If a patient does not agree to have the measurement following registration, the patient's registration on the study may be canceled. The Registrar should be notified of cancellations as soon as possible.

To register a patient, the following documents should be completed by the research nurse or data manager and faxed (336-713-6772) to the Registrar:

- Signed patient consent form/HIPAA authorization form
- On-Study/Registration Form (Appendix A)

The research nurse or data manager will then call (336-713-6767) the Registrar between the hours of 0800-1600 EST Monday-Friday to verify eligibility. To complete the registration process, the Registrar will:

- assign a patient study number
- register the patient on the study

### 7.0 Statistical Considerations

### Description of measures

### Standardized phase angle

Standardized phase angle will be calculated as in <sup>20</sup> (standardized phase angle = (measured phase angle–phase angle ref)/SD ref). Reference values and standard deviation come from measurements of phase angle in over 200,000 healthy German adults<sup>21</sup>.

### **Mortality**

30 day mortality rate is defined as the percent of patients no longer alive at 30 days after registration. In the rare case that a patient is lost to follow up before 30 days, the patient will be treated as missing.

60 day mortality rate is defined as the percent of patients no longer alive at 60 days after registration. Patients that are discharged to hospice care before 60 days without a known date of death will be counted towards 60 day mortality. In the rare case that a patient is lost to follow up before 60 days, the patient will be treated as missing.

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

### Treatment response

14 day bone marrow response is defined as hypoplastic marrow with less than 20% cellularity and 5% blasts.

Complete remission is defined as less than 5% marrow blasts, absolute neutrophil count >1000, platelet count >100,000 and freedom from red cell transfusions.

### Feasibility Analysis

If the study fails to accrue 20 patients during the first year of accrual it will be deemed unlikely to meet its ultimate accrual goal and the study will be terminated.

### Primary analysis

This study's primary endpoint is the association between standardized phase angle and 60 day mortality. Standardized phase angle will be treated as a continuous measure for the primary analysis. Since we will be using a standardized measure of phase angle, for power calculations we will assume a standard deviation of one and investigate the effects of a one unit change. A sample size of 102 patients would give us 80% power to detect an odds ratio of 2.1, using a logistic regression model with a 0.05 significance level and a 60 day mortality rate of 20%. With an expected accrual rate of 50 patients per year, the study should complete accrual in approximately two years and complete follow-up (two year follow-up) four years after the first patient is enrolled. Descriptive statistics will be used for baseline characteristics. Important baseline characteristics, such as age, will be added to the regression model as covariates for additional analysis.

### Secondary analysis

We will use logistic regression to analyze the association between standardized phase angle and the secondary outcomes of 30 day mortality, transfer to the intensive care unit, 14 day marrow response, complete remission and receipt of post-remission therapy. The association with overall survival will be evaluated using a Cox proportional hazards model. We will use a linear model to look at the association with length of hospital stay. It is likely that the length of hospital stay will not be normally distributed and will need a transformation to satisfy the normality assumption of the linear model. Feasibility will be analyzed qualitatively.

### Exploratory analysis

We will explore other versions of the standardized phase angle measure and how they relate to the primary and secondary outcomes. We will evaluate using categorical cut points of the baseline measure and the standardized phase angle measure captured just prior to the nadir marrow (for AML patients).

### 8.0 <u>Protection of Human Subjects</u>

Prior to implementation of this study, the protocol will be approved by the WFU Institutional Review Board (IRB). All subjects will provide written informed consent prior to enrollment in the study.

### 9.0 Data Submission Schedule

Appendix A – Eligibility Checklist and Registration Form:

- Submitted to Registrar at the time of registration

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

Appendix B – Demographics, Social and Medical History, Baseline Lab Data Collection Form:

- completed at study entry

### Appendix C – Comorbidity Data Collection Forms:

- completed at the time of initial phase angle measurement
- -submitted within one week of completion

### Appendix D – Phase Angle Measurement Form:

- completed each time a phase angle measurement is made (i.e. 1<sup>st</sup> day of treatment, prior to nadir marrow [AML patients only], and prior to any invasive procedures) -submitted within one week of completion

### Appendix E – Bone Marrow Biopsy and Treatment Data Collection Form:

- -completed as appropriate
- -submitted within one week of completion

### Appendix F – Follow-up Data Collection Form

- completed as appropriate
- -submitted within one week of completion

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

### 10.0 References

- 1. Licht JD, Sternberg DW. The molecular pathology of acute myeloid leukemia. *Hematology Am Soc Hematol Educ Program*. 2005:137-142. Prepublished on 2005/11/24 as DOI 2005/1/137 [pii]
- 10.1182/asheducation-2005.1.137.
- 2. Dohner H, Estey EH, Amadori S, et al. Diagnosis and management of acute myeloid leukemia in adults: recommendations from an international expert panel, on behalf of the European LeukemiaNet. *Blood*. 2010;115(3):453-474. Prepublished on 2009/11/03 as DOI blood-2009-07-235358 [pii]
- 10.1182/blood-2009-07-235358.
- 3. Siegel R, Ward E, Brawley O, Jemal A. Cancer statistics, 2011: The impact of eliminating socioeconomic and racial disparities on premature cancer deaths. *CA Cancer J Clin*. 2011;61(4):212-236. Prepublished on 2011/06/21 as DOI caac.20121 [pii] 10.3322/caac.20121.
- 4. Marks DI. Treating the "older" adult with acute lymphoblastic leukemia. *Hematology Am Soc Hematol Educ Program*. 2010;2010:13-20. Prepublished on 2011/01/18 as DOI 2010/1/13 [pii]
- 10.1182/asheducation-2010.1.13.
- 5. Larson RA. Treatment of older patients with acute lymphoblastic leukemia. *Annals of Hematology*. 2006;85:79-81.
- 6. Byrd JC, Mrozek K, Dodge RK, et al. Pretreatment cytogenetic abnormalities are predictive of induction success, cumulative incidence of relapse, and overall survival in adult patients with de novo acute myeloid leukemia: results from Cancer and Leukemia Group B (CALGB 8461). *Blood*. 2002;100(13):4325-4336. Prepublished on 2002/10/24 as DOI 10.1182/blood-2002-03-0772 [pii].
- 7. Rollig C, Thiede C, Gramatzki M, et al. A novel prognostic model in elderly patients with acute myeloid leukemia: results of 909 patients entered into the prospective AML96 trial. *Blood*. 2010;116(6):971-978. Prepublished on 2010/05/06 as DOI blood-2010-01-267302 [pii] 10.1182/blood-2010-01-267302.
- 8. Appelbaum FR, Gundacker H, Head DR, et al. Age and acute myeloid leukemia. *Blood*. 2006;107(9):3481-3485. Prepublished on 2006/02/04 as DOI 2005-09-3724 [pii] 10.1182/blood-2005-09-3724.
- 9. Brenner H, Pulte D, Gondos A. Improvement in survival in younger patients with acute lymphoblastic leukemia from the 1980s to the early 21st century. *Blood*. 2009;113(7):1408-1411. 10.1182/blood-2008-06-164863.
- 10. Juliusson G, Antunovic P, Derolf A, et al. Age and acute myeloid leukemia: real world data on decision to treat and outcomes from the Swedish Acute Leukemia Registry. *Blood*. 2009;113(18):4179-4187. Prepublished on 2008/11/15 as DOI blood-2008-07-172007 [pii] 10.1182/blood-2008-07-172007.
- 11. Kuendgen A, Germing U. Emerging treatment strategies for acute myeloid leukemia (AML) in the elderly. *Cancer Treat Rev.* 2009;35(2):97-120. Prepublished on 2008/10/28 as DOI S0305-7372(08)00284-3 [pii] 10.1016/j.ctrv.2008.09.001.

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

- 12. Larson RA. Acute lymphoblastic leukemia: older patients and newer drugs. *Hematology Am Soc Hematol Educ Program*. 2005:131-136. Prepublished on 2005/11/24 as DOI 2005/1/131 [pii]
- 10.1182/asheducation-2005.1.131.
- 13. Kantarjian H, Ravandi F, O'Brien S, et al. Intensive chemotherapy does not benefit most older patients (age 70 years or older) with acute myeloid leukemia. *Blood*. 2010. Prepublished on 2010/07/30 as DOI blood-2010-03-276485 [pii]
- 10.1182/blood-2010-03-276485.
- 14. Juliusson G. Older patients with acute myeloid leukemia benefit from intensive chemotherapy: an update from the Swedish Acute Leukemia Registry. *Clin Lymphoma Myeloma Leuk*. 2011;11 Suppl 1:S54-59. Prepublished on 2011/11/09 as DOI S2152-2650(11)00027-9 [pii]
- 10.1016/j.clml.2011.02.003.
- 15. Wheatley K, Brookes CL, Howman AJ, et al. Prognostic factor analysis of the survival of elderly patients with AML in the MRC AML11 and LRF AML14 trials. *Br J Haematol*. 2009;145(5):598-605. Prepublished on 2009/04/07 as DOI BJH7663 [pii] 10.1111/j.1365-2141.2009.07663.x.
- 16. Kyle UG, Bosaeus I, De Lorenzo AD, et al. Bioelectrical impedance analysis--part I: review of principles and methods. *Clin Nutr.* 2004;23(5):1226-1243. Prepublished on 2004/09/24 as DOI 10.1016/j.clnu.2004.06.004 S0261561404000937 [pii].
- 17. Faisy C, Rabbat A, Kouchakji B, Laaban JP. Bioelectrical impedance analysis in estimating nutritional status and outcome of patients with chronic obstructive pulmonary disease and acute respiratory failure. *Intensive Care Med.* 2000;26(5):518-525. Prepublished on 2000/08/03 as DOI.
- 18. Oliveira CM, Kubrusly M, Mota RS, Silva CA, Choukroun G, Oliveira VN. The phase angle and mass body cell as markers of nutritional status in hemodialysis patients. *J Ren Nutr*. 2010;20(5):314-320. Prepublished on 2010/03/23 as DOI S1051-2276(10)00009-9 [pii] 10.1053/j.jrn.2010.01.008.
- 19. Shah S, Whalen C, Kotler DP, et al. Severity of human immunodeficiency virus infection is associated with decreased phase angle, fat mass and body cell mass in adults with pulmonary tuberculosis infection in Uganda. *J Nutr*. 2001;131(11):2843-2847. Prepublished on 2001/11/06 as DOI.
- 20. Urbain P, Birlinger J, Ihorst G, Biesalski HK, Finke J, Bertz H. Body mass index and bioelectrical impedance phase angle as potentially modifiable nutritional markers are independent risk factors for outcome in allogeneic hematopoietic cell transplantation. *Ann Hematol.* 2013;92(1):111-119. Prepublished on 2012/09/13 as DOI 10.1007/s00277-012-1573-4.
- 21. Bosy-Westphal A, Danielzik S, Dorhofer RP, Later W, Wiese S, Muller MJ. Phase angle from bioelectrical impedance analysis: population reference values by age, sex, and body mass index. *JPEN J Parenter Enteral Nutr*. 2006;30(4):309-316. Prepublished on 2006/06/29 as DOI 30/4/309 [pii].

### Appendix A - Eligibility and Source Document Checklists, **Registration Form**

### CCCWFU # 99113

### **REGISTRATION GUIDELINES**

The following guidelines have been developed in order to ensure timely registration of your patient.

All patients entered on any CCCWFU trial, whether treatment, companion, or cancer control trial, **must** be registered with the CCCWFU Protocol Registrar or entered into ORIS Screening Log within 24 hours of Informed Consent. Patients must be registered prior to the initiation of treatment.

In order to ensure prompt registration of your patient, please:

- 1. Complete the Eligibility Checklist (attached)
- 2. Complete the Protocol Registration Form (attached)
- 3. Alert the WFUHS registrar by phone, and then send the signed Informed Consent Form, Eligibility Checklist and Protocol Registration Form to the registrar, either by fax or e-mail.

### Contact Information:

Protocol Registrar PHONE (336) 713-6767 Protocol Registrar FAX (336) 713-6772 Protocol Registrar E-MAIL (registra@wakehealth.edu)

\*Protocol Registration is open from 8:30 AM - 4:00 PM, Monday-Friday.

4. Please fax/e-mail ALL eligibility source documents with registration. Patients will **not** be registered without all required supporting documents.

Note: If labs were performed at an outside institution, please provide a printout of the results. Please ensure that the most recent lab values are sent.

CCCWFU # 99113

### **Eligibility Checklist**

Page 1

| Yes | No | N/A | Inclusion Criteria (All responses must be <b>YES</b> in order to enter study) | Eligibility<br>Confirmation<br>(registrar) |
|---|---|---|---|---|
| | | | <ol> <li>Is the patient hospitalized for newly diagnosed acute leukemia?</li> </ol> | |
| | | | <ol><li>Is the patient receiving induction treatment while hospitalized?</li></ol> | |
| | | | 3. Is the patient willing and able to provide written informed consent? | |
| Yes | No | N/A | Exclusion Criteria (All responses must be <b>NO</b> in order to enter | |
| | | | study) | |
| | | | <ol> <li>Does the patient have a pacemaker or defibrillator?</li> </ol> | |
| | | | 2. Is the patient pregnant? | |
| | | | 3. Does the patient have any abnormality which may, in the opinion of the investigator, compromise the safety of patients? | |
| | | | 4. Is the patient unable or unwilling to follow protocol requirements? | |

| Signature: | Date: |
|----------------------------------|---------------------------|
| Please send source documentation | on with Eligibility Form. |

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

CCCWFU # 99113

### Protocol Registration Form

Page 2

| DEMOGRAPHICS | |
|---|---|
| Patient: Last Name: | First Name: |
| MRN: | DOB (mm/dd/yy): / / |
| SEX: □ Male □ Female Ethnicity (choose one): □ Hispanic □Non | n-Hispanic |
| Race (choose all that apply): □ WHITE □BLACK □ ASIAN □ PA | ACIFIC ISLANDER |
| Height: inches | Weight:lbs.(actual) |
| Zip Code: | |
| Primary Diagnosis: | |
| Date of Diagnosis: / / | <del></del> |
| PROTOCOL INFORMATION | |
| Date of Registration: | // |
| MD Name (last) : | <del></del> |
| Informed written consent (consent must be ☐ YES ☐ NO | signed prior to registration): |
| Date Consent Signed: | / |
| PID # (to be assigned by ORIS): | |

Protocol Registrar can be contact by calling 336-713-6767 between 8:30 AM and 4:00 PM, Monday — Friday. Completed Eligibility Checklist and Protocol Registration Form must be hand delivered, faxed or e-mailed to the registrar at 336-7136772 or registra@wakehealth.edu.

## CCCWFU # 99113 Eligibility Source Documentation Checklist Page 3 (to be submitted with Protocol Registration Form)

| | Source Documents Needed | √ or<br>N/A |
|---|---|---|
| 1 | Documentation that patient is hospitalized for newly diagnosed acute leukemia | |
| 2 | Documentation that patient is receiving induction treatment while hospitalized | |
| 3 | Signed informed consent document | |
| 4 | Documentation that patient is not pregnant | |
| 5 | Documentation that patient is free from any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients | |

### Appendix B: Social and Medical History, Baseline Lab Data Collection Form 

| Demographics<br>Social History: | | | |
|---|---|---|---|
| Married: | Yes No _ | | |
| Tobacco use: | Current | Former | Never |
| Alcohol abuse: | Current | Former | Never |
| Baseline Labs on<br>WBC<br>HEMOGLOBIN<br>HEMATOCRIT | date of admissior | SODIUM<br>POTASSIUM<br>BUN | mal point)<br> |
| PLATELETS<br>NEUTROPHILS<br>BANDs<br>ANC | | GLUCOSE<br>CREATININE<br>ALBUMIN<br>T. BILIRUBIN<br>ALK PHOS<br>AST | |
| LDH | · | AST<br>ALT<br>GFR | |

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

## Appendix B: Demographics, Social and Medical History, Baseline Lab Data Collection Form 

### **Past Medical History** Number of comorbidities: (0-20) Past History of: (per documentation in medical record at time of admission) Congestive Heart Failure Y N Depression Y\_\_\_ N\_\_\_ Coronary artery disease Y N Osteoporosis Y N Y \_ N\_\_\_ Cerebrovascular Disease Y N Rheumatologic disease (SLE, RA, scleroderma, Sjogrens) (Stroke, TIA) Y \_ N\_\_\_ Diabetes Mellitus Y N Cognitive Impairment Y\_\_\_ N\_\_\_ COPD VTE (Venous thrombosis, DVT, PE) (Emphysema) Hypertension Y N Cardiac valve disease Y \_ N\_\_\_ Y\_\_\_ N\_\_\_ Y\_\_\_ N\_\_\_ Renal Dysfunction Cirrhosis (Excludes non-melanoma skin) Y\_\_\_N\_\_\_ MDS (H&P only) MDS (path report only) Y\_\_\_N\_\_ If yes, then cancer type \_\_\_\_\_ Prior treatment with: (check) Chemotherapy \_\_\_\_ Radiation \_\_\_\_ Surgery \_\_\_\_

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

### **Appendix C: Comorbidity Data Collection Forms **

### **Charlson Comorbidity Index**

### Comorbidity and score (circle) Myocardial infarction 1 **Congestive heart failure** 1 Cerebrovascular disease 1 Peptic ulcer 1 Hepatic ulcer (mild) 1 **Diabetes** (mild/moderate) 1 **Pulmonary disease** (mild/moderate) 1 **Diabetes** (with severe end stage organ damage) 2 2 Renal disease (moderate or severe) **Hepatic disease** (moderate or severe) 3 Solid tumor with metastases 6 Total Score\_\_\_\_

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

### **Appendix C: Comorbidity Data Collection Forms **

### Hematopoietic Cell Transplant Comorbidity Index (HCT-CI)

| ricinatopoletic och fransplant comorbiatty mack | (1101-0 |
|---|---|
| Comorbidity and score (circle) | |
| Cardiac<br>(CAD, CHF, MI, EF ≤ 50%) | 1 |
| Arrhythmia (Atrial fibrillation or flutter, sick sinus or ventricular arrhythmia) | 1 |
| Cerebrovascular disease<br>(TIA or CVA) | 1 |
| Peptic ulcer<br>(Requiring treatment) | 2 |
| Hepatic Disease (mild) (Chronic hepatitis, bilirubin>ULN to 1.5 X the ULN,or AST/ALT>ULN to 2.5 X the ULN) | 1 |
| <b>Diabetes</b> (Requiring treatment with medication) | 1 |
| Pulmonary (moderate) (DLCO and/or FEVI 66-80% or dyspnea with slight activity) | 2 |
| Rheumatologic<br>(SLE, RA, polymyositis, mixed CTD,<br>or polymyalgia rheumatica) | 2 |
| Inflammatory bowel disease<br>(Crohns disease or ulcerative colitis) | 1 |
| Renal (moderate/severe) (Serum creatinine>2mg/dL, mixed CTD, or prior renal transplant) | 2 |
| Prior solid tumor<br>(Treated at any point in patient's history,<br>excluding non-melanoma) | 3 |

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

### **Appendix C: Comorbidity Data Collection Forms **

| Total scor | e: |
|---|---|
| Severe pulmonary<br>(DLCO and or FEVI ≤ 65% or dyspnea at rest or requiring oxyger | 3 |
| Heart Valve Disease<br>(Except mitral valve prolapse) | 3 |
| Psychiatric Disturbance (Depression or anxiety requiring psychiatric consult or treatment) | 1 |
| Infection (Requiring use of antimicrobial treatment) | 1 |
| <b>Obesity</b> (Body mass index > 35 kg/m²) | 1 |
| <b>Hepatic</b> (moderate/severe) (Liver cirrhosis, bilirubin>1.5 X the ULN, or AST/ALT>2.5 X the ULN) | 3 |

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

### **Appendix D – Phase Angle Measurement Form**

To be completed with each phase angle measurement:

| ORIS Assigned PID: |
|---|
| Physical Exam: |
| Date of Exam: / / |
| Weight: (kg) |
| Height: (cm) |
| Systolic Blood Pressure (SBP): (50-250) |
| Diastolic Blood Pressure (DBP): (30-130) |
| Pulse: (30-180) |
| Phase Angle: R: Xc |
| For AML Patients: Second Phase Angle Measurement taken just prior to the nadir marrow <a href="Physical Exam">Physical Exam</a> : |
| Date of Exam: / / |
| Weight: (kg) |
| Height: (cm) |
| Systolic Blood Pressure (SBP): (50-250) |
| Diastolic Blood Pressure (DBP): (30-130) |
| Pulse: (30-180) |
| Phase Angle: |

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

### **Appendix E – Bone Marrow Biopsy and Treatment Data Collection Forms**

| BONE MARROW BIOPSY: |
|---|
| DATE/ |
| Diagnosis: AML or ALL Blast %: |
| CYTOGENETICS:(free text) |
| RISK GROUP: FAVORABLE INTERMEDIATE UNFAVORABLE |
| APL: YES NO Hypoplastic marrow cellularity %: |
| TREATMENT: |
| HOSPITALIZED FOR INDUCTION CHEMOTHERAPY: Y N |
| DATE OF ADMISSION: |
| DATE OF DISCHARGE: |
| DATE INDUCTION CHEMOTHERAPY INITIATED: |
| TYPE OF CHEMOTHERAPY ADMINISTERED (check one): |
| <ol> <li>AraC+anthracycline+etoposide (7+3+3)</li> <li>AraC+ anthracycline (7+3)</li> <li>As per CALGB 10102</li> <li>other</li></ol> |
| NUMBER OF CYCLES OF CHEMOTHERAPY:(range 0-5) |
| RESIDUAL DISEASE ON 14-DAY BONE MARROW BIOPSY: Y N N/A |
| REQUIRED ICU DURING HOSPITAL STAY: Y N |
| DEATH WITHIN 30 DAYS OF INITIAL TREATMENT: Y N |
| DEATH WITHIN 60 DAYS OF INITIAL TREATMENT: Y N |
| DISPOSITION: HOME SNFALF HOSPICE DECEASED |
| Need for total parenteral nutrition or feeding tube placement during induction hospitalization: |
| Y N |

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

## Appendix F -FOLLOW-UP (POST INDUCTION HOSPITALIZATION) Data Collection Form 

| COMPLETE REMISS Comment for Complete Remissio RECEIVED POST-REMISSION T Number of cycles of consolidation | n:(free text, 200 characters) THERAPY: Y N |
|---|---|
| Complete consolidation informati | on below as applicable: |
| Date of 1 <sup>st</sup> consolidation: | |
| Specify type of 1 <sup>st</sup> consolidation: | hypomethylating agent (5-azacitidine/decitabine) |
| | autologous transplantation |
| | reduced intensity allogeneic transplant |
| | full allogeneic transplant |
| | Ara-C |
| | If received Ara-C for 1 <sup>st</sup> consolidation, record dose: 3gm/m <sup>2</sup> 2 gm/m <sup>2</sup> 1.5 g/m <sup>2</sup> 1gm/m <sup>2</sup> 500mg/m <sup>2</sup> |
| | Other |
| Date of 2 <sup>nd</sup> consolidation: | If other record type:(text, 50 characters) |
| | hypomethylating agent (decitabine/azacitidine) |
| | autologous transplantation |
| | reduced intensity allogeneic transplant |
| | full allogeneic transplant |
| | Ara-C |
| | If received Ara-C for 2 <sup>nd</sup> consolidation, record dose: 3gm/m <sup>2</sup> 2 gm/m <sup>2</sup> 1.5 g/m <sup>2</sup> 1gm/m <sup>2</sup> 500mg/m <sup>2</sup> |
| | Other |
| | If other record type:(text, 50 characters) |
| | (text, 50 Glaracters) |

## CCCWFU #99113 – Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia

## Appendix F -FOLLOW-UP (POST INDUCTION HOSPITALIZATION) Data Collection Form 

| Date of 3 <sup>rd</sup> consolidation: | <del></del> |
|---|---|
| Specify type of 3 <sup>rd</sup> consolidation: | hypomethylating agent (decitabine/azacitidine) |
| | autologous transplantation |
| | reduced intensity allogeneic transplant |
| | full allogeneic transplant |
| | Ara-C |
| | If received Ara-C for 3 <sup>rd</sup> consolidation, record dose: 3gm/m <sup>2</sup> 2 gm/m <sup>2</sup> 1.5 g/m <sup>2</sup> 1gm/m <sup>2</sup> 500mg/m <sup>2</sup> |
| | Other |
| | If other record type: (text, 50 characters) |
| RECEIVED BONE MARROW TRA | ANSPLANTATION: Y N |
| IF YES, SPECIFY TYPE: (PICK ( | ONE) REDUCED INTENSITY<br>FULL ALLOGENEIC<br>AUTOLOGOUS |
| SPECIFY REGIMEN: | (FREE TEXT, 100 characters) |
| Date of bone marrow transplant: | |

| Appendix G – Survival Data |
|-------------------------------------------------|
| ORIS Assigned PID: |
| Visit Date: / / |
| Visit Interval: |
| 3 Mos Post 6 Mos Post 9 Mos Post 12 Mos Post |
| 15 Mos Post 18 Mos Post 21 Mos Post 24 Mos Post |
| Other Mos Post Number of Months Post Discharge |
| DATE OF LAST CONTACT: / / |
| <b>DECEASED</b> : Y N |
| DATE OF DEATH: / / |